CLINICAL TRIAL: NCT00549302
Title: An Extension Study to Evaluate the Long-Term Safety and Efficacy of the Phosphodiesterase Type 5 (PDE5) Inhibitor Tadalafil in the Treatment of Patients With Pulmonary Arterial Hypertension
Brief Title: Study the Safety and Effectiveness of Tadalafil on High Blood Pressure in the Blood Vessel Going From the Heart to the Lungs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ICOS Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10263; H6D-MC-LVGX (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-10-23; First posted 2007-10-25 (Estimated); Results first posted 2013-02-18 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Hypertension, Pulmonary
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 20 mg tadalafil (Active Comparator): 20 milligram (mg) tadalafil taken once a day
  Interventions: Drug: tadalafil
- 40 mg tadalafil (Active Comparator): 40 mg tadalafil tablet taken once a day
  Interventions: Drug: tadalafil

INTERVENTIONS:
Drug: tadalafil — 20 milligram (mg) tablet, taken by mouth once a day for 52 weeks for the phase 1 portion. Open label phase includes 40 mg tablet taken by mouth once a day until the sponsor concludes the study or tadalafil becomes commercially available for the treatment of Pulmonary Arterial Hypertension (PAH).
  Other Names: LY450190; Cialis; IC351
  Arms: 20 mg tadalafil
Drug: tadalafil — 40 mg tablet taken by mouth once a day for 52 weeks in phase 1. Open label phase includes 40 mg tablet taken by mouth once a day until the sponsor concludes the study or tadalafil becomes commercially available for the treatment of PAH.
  Other Names: LY450190; Cialis; IC351
  Arms: 40 mg tadalafil

SUMMARY:
Study to determine the long term safety of tadalafil in patients with increased blood pressure in the blood vessel that carries blood from the right heart to the lungs and to see if it will keep the disease from getting worse.

ELIGIBILITY:
Inclusion Criteria:

* Must have participated and discontinued in the previous PAH placebo controlled study due to clinical worsening on placebo or tadalafil 2.5 mg, 10mg, or 20 mg
* Must have completed Week 16 of the previous PAH study and had either no clinical worsening or became clinically worse at the Week 16 visit on placebo or tadalafil 2.5 mg, 10mg, or 20 mg
* Females who have a negative urine pregnancy test and are willing to use 2 types of birth control
* Be 12 years or older (country specific regulations apply) with parental approval

Exclusion Criteria:

* Participated in the placebo controlled study and had clinical worsening on 40 mg tadalafil
* Have left-sided heart disease
* Have a musculoskeletal disorder that limits being able to get around
* Nitrate use
* Certain current systemic treatments

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2005-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (10):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon- Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bend, Oregon, United States
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon- Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brussels, Belgium
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon- Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario, Canada
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon- Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille, France
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon- Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin, Germany
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon- Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dublin, Ireland
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon- Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bergamo, Italy
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon- Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo, Japan
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon- Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona, Spain
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon- Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, United Kingdom

REFERENCES:
- [Derived] Oudiz RJ, Brundage BH, Galie N, Ghofrani HA, Simonneau G, Botros FT, Chan M, Beardsworth A, Barst RJ; PHIRST Study Group. Tadalafil for the treatment of pulmonary arterial hypertension: a double-blind 52-week uncontrolled extension study. J Am Coll Cardiol. 2012 Aug 21;60(8):768-74. doi: 10.1016/j.jacc.2012.05.004. Epub 2012 Jul 18. PMID 22818063
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were previously enrolled in H6D-MC-LVGY (NCT00125918), a placebo-controlled double-blind study.
Groups:
- Tadalafil 20 mg Double Blind: Tadalafil, 20 milligram (mg) administered orally as 1 tadalafil tablet and 1 matched placebo tablet once daily from Day 1 up to 52 weeks of treatment.
- Tadalafil 40 mg Double-Blind: Tadalafil, 40 mg (two 20 mg tablets) administered orally once daily from Day 1 up to 52 weeks of treatment.
- Tadalafil 40 mg Open-Label: Tadalafil, 40 mg (two 20 mg tablets) administered orally once daily from Week 53 up to Week 243.
Period: Double-Blind
Arm/Group | Tadalafil 20 mg Double Blind | Tadalafil 40 mg Double-Blind | Tadalafil 40 mg Open-Label
Started | 63 | 294 | 0
Received at Least One Dose of Study Drug | 63 | 294 | 0
Completed | 52 (Participants who completed the Double-Blind Period were eligible to enter the Open-Label Period.) | 241 (Participants who completed the Double-Blind Period were eligible to enter the Open-Label Period.) | 0
Not Completed | 11 | 53 | 0
Not completed — Death | 2 | 9 | 0
Not completed — Adverse Event | 3 | 16 | 0
Not completed — Withdrawal by Subject | 3 | 8 | 0
Not completed — Investigator Decision | 1 | 5 | 0
Not completed — Sponsor Decision | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0
Not completed — New Drug Pulmonary Atrial Hypertension | 1 | 10 | 0
Not completed — New condition or starts new therapy | 0 | 2 | 0
Period: Open-Label
Arm/Group | Tadalafil 20 mg Double Blind | Tadalafil 40 mg Double-Blind | Tadalafil 40 mg Open-Label
Started | 0 | 0 | 286 (7 participants who completed the Double-Blind Period did not enter the Open-Label Period.)
Completed | 0 | 0 | 217 (Another death occurred during the 30-day follow-up period after study drug discontinuation)
Not Completed | 0 | 0 | 69
Not completed — Adverse Event | 0 | 0 | 11
Not completed — Death | 0 | 0 | 40
Not completed — Investigator Decision | 0 | 0 | 5
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Other | 0 | 0 | 3
Not completed — New drug pulmonary atrial hypertension | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Tadalafil 20 Milligrams (mg) Double-Blind: Tadalafil, 20 milligram (mg) administered orally as 1 tadalafil tablet and 1 matched placebo tablet once daily from Day 1 up to 52 weeks of treatment.
- Total: Total of all reporting groups
Arm/Group | Tadalafil 20 Milligrams (mg) Double-Blind | Tadalafil 40 mg Double-Blind | Total
Number analyzed (Participants) | 63 | 294 | 357
Age Continuous [Mean (Standard Deviation); unit: years] | 53.04 (15.58) | 53.94 (15.36) | 53.78 (15.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 230 | 278
  Male | 15 | 64 | 79
Region of Enrollment [Number; unit: participants]
  Belgium | 2 | 5 | 7
  Canada | 4 | 38 | 42
  France | 3 | 22 | 25
  Germany | 6 | 34 | 40
  Ireland | 0 | 1 | 1
  Italy | 4 | 25 | 29
  Japan | 5 | 17 | 22
  Spain | 2 | 4 | 6
  United States | 33 | 139 | 172
  United Kingdom | 4 | 9 | 13
Race [Number; unit: participants]
  White | 48 | 243 | 291
  Asian | 7 | 22 | 29
  Black or African American | 5 | 23 | 28
  American Indian or Alaska Native | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  American Indian or Alaska Native/White | 0 | 1 | 1
  Black or African American/Native Hawaiian or Other | 1 | 0 | 1
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 73.92 (18.90) | 75.26 (19.80) | 75.02 (19.63)
Ethnicity [Number; unit: participants]
  Hispanic or Latino | 4 | 36 | 40
  Not Hispanic or Latino | 59 | 258 | 317
Etiology [Number; unit: participants]
  Idiopathic | 37 | 186 | 223
  Related to Collagen Vascular Disease | 16 | 62 | 78
  Associated with Atrial Septal Defect | 3 | 26 | 29
  Related to Anorexigen Use | 4 | 11 | 15
  Surgical Repair, of at least 1 Year Duration | 3 | 9 | 12
Current Bosentan Use [Number; unit: participants]
  Yes | 37 | 155 | 192
  No | 26 | 139 | 165

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: A summary of serious and all other non-serious AEs, which include adverse events reported for laboratory tests and vital signs, is located in the Reported Adverse Event module.
Time Frame: Baseline (Double-Blind Period) up to Week 243 (End of Open-Label Period)
Population: Safety Population: all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Groups:
- Tadalafil 20 mg or 40 mg Double-Blind and 40 mg Open-Label: Tadalafil 20 mg tablets administered orally as one tablet tadalafil and one tablet matched placebo once per day from Day 1 up to 52 weeks of treatment or tadalafil, two 20 mg tablets (40 mg total) administered orally once per day from Day 1 up to 52 weeks of treatment in Double-blind period; and tadalafil, two 20 mg tablets (40 mg total) administered orally once per day from Week 53 up to Week 243 in Open-label period.
Arm/Group | Tadalafil 20 mg or 40 mg Double-Blind and 40 mg Open-Label
Number analyzed (Participants) | 357
participants
  Serious AEs | 184
  Other Non-Serious AEs | 334

2. Secondary Outcome: 6-Minute Walk Distance (6MWD) at Baseline and Weeks 16, 28, 40 and 52
Description: 6MWD measured the distance a participant was able to walk unassisted in 6 minutes.
Time Frame: Baseline and Weeks 16, 28, 40 and 52
Population: All randomized participants who received at least 1 dose of study drug and who completed 6MWD test; Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: meters (m)
Arm/Group | Tadalafil 20 Milligrams (mg) Double-Blind | Tadalafil 40 mg Double-Blind
Number analyzed (Participants) | 63 | 284
meters (m)
  Distance walked at Baseline (n=63, 287 | 397.74 (71.74) | 375.38 (93.41)
  Distance walked at Week 16 (n=58, 272) | 396.37 (77.01) | 381.47 (96.86)
  Distance walked at Week 28 (n=55, 250) | 406.41 (106.76) | 384.97 (95.03)
  Distance walked at Week 40 (n=51, 241) | 411.81 (78.72) | 386.57 (94.04)
  Distance walked at Week 52 (n=51, 235) | 415.31 (79.82) | 394.00 (91.56)
  Endpoint-Week 52 or LOCF (n=60,281) | 401.52 (90.29) | 379.80 (99.12)

3. Secondary Outcome: Borg Dyspnea Assessment at Baseline and Weeks 16, 28, 40 and 52
Description: Borg dyspnea score is a participant rated measure of their greatest degree of shortness of breath during exertion (6-minute walk test). Score ranged from 0 (nothing at all) to 10 (very, very severe [maximal]).
Time Frame: Baseline and Weeks 16, 28, 40 and 52
Population: All randomized participants who received at least 1 dose of study drug and who completed the Borg Dyspnea Assessment; LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tadalalfil 20 Milligrams (mg): Tadalafil, 20 milligram (mg) tablets administered orally as one tablet tadalafil and one tablet matched placebo once per day from Day 1 up to 52 weeks of treatment; LOCF.
- Tadalafil 40 mg: Tadalafil, two 20 mg tablets (40 mg total) administered orally once per day from Day 1 up to 52 weeks of treatment.
Arm/Group | Tadalalfil 20 Milligrams (mg) | Tadalafil 40 mg
Number analyzed (Participants) | 63 | 294
units on a scale
  Score at Baseline (n=62, 287) | 3.41 (2.38) | 3.65 (2.43)
  Score at Week 16 (n=58, 271) | 3.41 (2.48) | 3.51 (2.35)
  Score at Week 28 (n=54,249) | 3.46 (2.40) | 3.44 (2.21)
  Score at Week 40 (n=51, 240) | 3.21 (2.43) | 3.38 (2.27)
  Score at Week 52 (n=51,235) | 3.68 (2.43) | 3.29 (2.16)
  Endpoint-Week 52 or LOCF (n=60,281) | 3.75 (2.34) | 3.54 (2.36)

4. Secondary Outcome: Probability of No Pulmonary Arterial Hypertension (PAH) Deterioration at Weeks 16, 28, 40 and up to 52
Description: World Health Organization Functional Classification Assessment (WHO FC) is a method of classifying disease severity in PAH. The classes are: Class I: pulmonary hypertension (PH) but without resulting limitation of physical activity, Class II: PH resulting in slight limitation of physical activity, Class III: PH resulting in marked limitation of physical activity, Class IV: PH with inability to carry out any physical activity without symptoms. Deterioration of WHO FC is defined as moving to a higher WHO FC within one visit. Results are presented as Kaplan-Meier estimates (% probability) of remaining free from WHO FC deterioration after a given time.
Time Frame: Baseline and Weeks 16, 28, 40 and 52
Population: Safety Population: all randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: probability (%) no PAH deterioration
Arm/Group | Tadalafil 20 Milligrams (mg) Double-Blind | Tadalafil 40 mg Double-Blind
Number analyzed (Participants) | 63 | 294
probability (%) no PAH deterioration
  Week 16 (n=57, 262) | 95 [85 to 98] | 96 [93 to 98]
  Week 28 (n=50, 238) | 88 [77 to 94] | 90 [86 to 93]
  Week 40 (n=45, 222) | 81 [68 to 89] | 88 [83 to 91]
  Week 52 (n=33,136) | 81 [68 to 89] | 85 [80 to 89]

ADVERSE EVENTS:
Description: All treatment emergent adverse events (TEAEs) defined as a Serious Adverse Event (SAEs) and Other Non-serious Adverse Event (AEs) which were either first reported or worsened in severity during the Double-Blind Period or the Open-Label Period when compared with baseline observed in Study LVGY (NCT00125918) and were merged into 1 reporting group.
Groups:
- Tadalafil 20 mg or 40 mg Double-Blind and 40 mg Open-Label: Tadalafil 20 mg administered orally as 1 tadalafil 20-mg tablet and 1 matched placebo tablet, once daily from Day 1 up to 52 weeks of treatment, or tadalafil 40 mg (two 20-mg tablets) administered orally, once daily from Day 1 up to 52 weeks of treatment in Double-Blind Period; and tadalafil 40 mg (two 20-mg tablets) administered orally, once daily from Week 53 up to Week 243 in Open-Label Period.
Arm/Group | Tadalafil 20 mg or 40 mg Double-Blind and 40 mg Open-Label
Serious Adverse Events (participants affected / at risk) | 184/357
Other Adverse Events (participants affected / at risk) | 334/357
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil 20 mg or 40 mg Double-Blind and 40 mg Open-Label (N=357)
Anaemia (Blood and lymphatic system disorders) | 7 (11)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2)
Angina pectoris (Cardiac disorders) | 3 (3)
Angina unstable (Cardiac disorders) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1) — Resulted in 1 participant death in the Tadalafil 40 mg open-label arm
Arrhythmia (Cardiac disorders) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 7 (11)
Atrial flutter (Cardiac disorders) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 5 (5) — Resulted in 3 participant deaths, 1 in the Tadalafil 40 mg arm and 2 in the Tadalafil 40 mg open-label arm
Cardiac failure (Cardiac disorders) | 9 (10) — Resulted in 5 participant deaths 4 in the Tadalafil 40 mg open-label arm and 1 in the 30-day follow-up period after study drug discontinuation
Cardiac failure congestive (Cardiac disorders) | 10 (16) — Resulted in 3 participant deaths in the Tadalafil 40 mg open-label arm
Cardiac flutter (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) — Resulted in 1 participant death in the Tadalafil 40 mg open-label arm
Cardio-respiratory distress (Cardiac disorders) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) — Resulted in 1 participant death in the Tadalafil 40 mg open-label arm
Cor pulmonale (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2)
Cyanosis (Cardiac disorders) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 4 (5) — Resulted in 3 participant deaths, 1 death in the Tadalafil 40 mg and 2 in the Tadalafil 40 mg open-label arm
Palpitations (Cardiac disorders) | 3 (3)
Pericardial haemorrhage (Cardiac disorders) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 1 (1)
Right ventricular failure (Cardiac disorders) | 28 (36) — Resulted in 9 participant deaths, 2 in the Tadalafil 40 mg arm and 7 in the Tadalafil 40 mg open-label arm
Sick sinus syndrome (Cardiac disorders) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 3 (3)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Visual disturbance (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1)
Colonic polyp (Gastrointestinal disorders) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastric volvulus (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 (10)
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 (1)
Gingival hypertrophy (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (2)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Intestinal polyp (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Oesophageal achalasia (Gastrointestinal disorders) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Chest pain (General disorders) | 7 (9)
Chills (General disorders) | 1 (1)
Cyst (General disorders) | 1 (1)
Death (General disorders) | 3 (3) — Resulted in 3 participant deaths, 1 in the Tadalafil 40 mg arm and 2 in the Tadalafil 40 mg open-label arm
Device malfunction (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Injection site haemorrhage (General disorders) | 1 (1)
Medical device complication (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 4 (4)
Oedema peripheral (General disorders) | 5 (5)
Pyrexia (General disorders) | 3 (4)
Sensation of pressure (General disorders) | 1 (1)
Sudden cardiac death (General disorders) | 2 (2) — Resulted in 2 participant deaths in the Tadalafil 40 mg arm
Sudden death (General disorders) | 2 (2) — Resulted in 2 participant deaths, 1 in the Tadalafil 20 mg arm and another in the Tadalafil 40 mg open-label arm
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 2 (2)
Bronchiolitis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 6 (6)
Bronchitis bacterial (Infections and infestations) | 1 (1)
Campylobacter infection (Infections and infestations) | 1 (1)
Campylobacter intestinal infection (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Clostridial infection (Infections and infestations) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 2 (2)
Device related infection (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Herpes zoster ophthalmic (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 2 (2)
Lobar pneumonia (Infections and infestations) | 1 (1) — Resulted in 1 participant death in the Tadalafil 40 mg open-label arm
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 3 (3) — Resulted in 1 participant death in the Tadalafil 40 mg open-label arm
Mycobacterial infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (2)
Parotitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 16 (19) — Resulted in 2 participant deaths, 1 in the Tadalafil 40 mg arm and another death in the Tadalafil 40 mg open-label arm
Pneumonia staphylococcal (Infections and infestations) | 1 (1) — Resulted in 1 participant death in the Tadalafil 40 mg open-label arm
Pulmonary tuberculosis (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Septic shock (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 2 (2)
Staphylococcal skin infection (Infections and infestations) | 2 (2)
Tracheobronchitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (3)
Viral infection (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (5)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 2 (2)
Post procedural discharge (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1)
Pubic rami fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 (3)
Blood pressure increased (Investigations) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1)
Cardiac output decreased (Investigations) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 6 (6)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 4 (5)
Fluid retention (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bunion (Musculoskeletal and connective tissue disorders) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2)
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (3)
Systemic sclerosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Leiomyosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Resulted in 1 participant death in the Tadalafil 40 mg open-label arm
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Resulted in 1 participant death in the Tadalafil 40 mg arm
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) — Resulted in 1 participant death in the Tadalafil 40 mg open-label arm
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Resulted in 1 participant death in the Tadalafil 40 mg open-label arm
Oropharyngeal cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Uterine leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Cervical myelopathy (Nervous system disorders) | 1 (1)
Complicated migraine (Nervous system disorders) | 1 (1)
Dementia (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Dystonia (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 10 (10)
Transient ischaemic attack (Nervous system disorders) | 2 (2)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 1 (2)
Bipolar disorder (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Emotional disorder (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 2 (2)
Withdrawal syndrome (Psychiatric disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 5 (7)
Renal failure chronic (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Resulted in 1 participant death in the Tadalafil 40 mg open-label arm
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Resulted in 1 participant death in the Tadalafil 40 mg open-label arm
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 26 (28) — Resulted in 3 participant deaths in the Tadalafil 40 mg open-label arm
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6) — Resulted in 4 participant deaths in the Tadalafil 40 mg open-label arm
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 (3)
Skin lesion excision (Surgical and medical procedures) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) — Resulted in 1 participant death in the Tadalafil 40 mg arm
Haematoma (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Hypertensive crisis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Paradoxical embolism (Vascular disorders) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil 20 mg or 40 mg Double-Blind and 40 mg Open-Label (N=357)
Anaemia (Blood and lymphatic system disorders) | 42 (51)
Palpitations (Cardiac disorders) | 52 (61)
Vision blurred (Eye disorders) | 22 (23)
Diarrhoea (Gastrointestinal disorders) | 77 (107)
Dyspepsia (Gastrointestinal disorders) | 35 (39)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 19 (19)
Nausea (Gastrointestinal disorders) | 44 (56)
Vomiting (Gastrointestinal disorders) | 18 (22)
Asthenia (General disorders) | 18 (18)
Chest pain (General disorders) | 38 (45)
Fatigue (General disorders) | 49 (56)
Oedema peripheral (General disorders) | 63 (82)
Bronchitis (Infections and infestations) | 34 (44)
Influenza (Infections and infestations) | 26 (31)
Nasopharyngitis (Infections and infestations) | 64 (110)
Respiratory tract infection (Infections and infestations) | 19 (30)
Sinusitis (Infections and infestations) | 27 (42)
Upper respiratory tract infection (Infections and infestations) | 63 (105)
Urinary tract infection (Infections and infestations) | 37 (59)
Hypokalaemia (Metabolism and nutrition disorders) | 20 (25)
Arthralgia (Musculoskeletal and connective tissue disorders) | 40 (43)
Back pain (Musculoskeletal and connective tissue disorders) | 64 (76)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 29 (31)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 19 (19)
Myalgia (Musculoskeletal and connective tissue disorders) | 28 (30)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 44 (51)
Dizziness (Nervous system disorders) | 61 (73)
Headache (Nervous system disorders) | 107 (130)
Syncope (Nervous system disorders) | 20 (25)
Anxiety (Psychiatric disorders) | 23 (24)
Depression (Psychiatric disorders) | 22 (25)
Insomnia (Psychiatric disorders) | 36 (37)
Cough (Respiratory, thoracic and mediastinal disorders) | 54 (61)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 55 (69)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 39 (44)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 27 (31)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 33 (41)
Rash (Skin and subcutaneous tissue disorders) | 29 (32)
Flushing (Vascular disorders) | 28 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days